CLINICAL TRIAL: NCT02842138
Title: A Safety and Efficacy Study of Autologous T Cells Engineered to Express Chimeric Antigen Receptor Targeting CD19 in Patients With Relapsed or Refractory B-cell Lymphoma
Brief Title: Autologous CD19 CAR T Cells in Relapsed or Refractory B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Collaborators: Marino Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhu, Principal Investigator, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016YJZ12
Record Dates: First submitted 2016-07-13; First posted 2016-07-22 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD19 CAR T cells (Experimental): A standard dose escalation approach aimed to assess the safety and efficacy of autologous anti-CD19 CAR T cells will be applied.
  Interventions: Biological: autologous anti-CD19 CAR T cells

INTERVENTIONS:
Biological: autologous anti-CD19 CAR T cells — Patients will receive a three-day regimen of chemotherapy consisting of fludarabine and cyclophosphamide aimed to deplete the lymphocytes. Four days after lymphodepletion, patients are intravenously infused autologous anti-CD19 CAR T cells. A prescribed CAR T cell dose will be intravenously infused to patient in a three-day split-dose regimen (day0,30%; day1, 30%; day2, 40%).

SUMMARY:
This is a single arm, open-label, one center, dose escalation clinical study to determine the safety and efficacy of infusion of autologous T cells expressing CD19-redirected Chimeric Antigen Receptor (CD19 CAR T) in adult patients with relapsed or refractory CD19 positive B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. CD19+ B cell lymphoma,verified by IHC or flow cytometry.
2. a prior history of at least two standard care of medication.
3. ineligible for allogeneic transplantation or relapsed after transplantation.
4. patients are 18 years older.
5. life expectancy > 3months.
6. ECOG ≤ 2.
7. satisfactory major organ functions: adequate heart function with LVEF≥50%; pulse oximetry of ≥ 90%; cockcroft-gault creatinine clearance≥40 ml/min; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3ULN; Bilirubin ≤2.0 mg/dl .
8. Blood: Hgb ≥ 80 g/L, ANC ≥ 1×10^9/L, PLT ≥ 50×10^9/L.
9. women of reproductive potential must have a negative pregnancy test. Male and female of reproductive potential must agree to use birth control during the study and one year post study.
10. measurable tumors.

Exclusion Criteria:

1. using immunosuppressive drugs or systemic steroids within one week of enrollment.
2. active infection.
3. HIV positive.
4. active hepatitis B virus infection or hepatitis C virus infection.
5. breastfeeding or pregnant women.
6. patients refuse to practice birth control during study and one year post study.
7. patients with a prior history of other malignances will be excluded from this study, but patients who have been cured from skin basal cell carcinoma or cervical cancer, or who have had their tumors removed by surgical resection but without further therapies and have more than 5 years of progression-free survival, can be included into the study.
8. currently enrolled in other study.
9. patients, in the opinion of investigators, may not be eligible or are not able to comply with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-02-28 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 2 years

SECONDARY OUTCOMES:
Treatment response rate of anti-CD19 CAR T cell infusion | 4 weeks
  Defined as the proportion of patients who achieved complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD) based on standardized response criteria for malignant lymphoma (Cheson BD, JCO, 2007).
overall survival rate of patients treated with anti-CD19 CAR T cells | 2 years
progression-free survival of patients treated with anti-CD19 CAR T cells | 2 years

OTHER OUTCOMES:
Persistence of CAR T cells in patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ying Z, Huang XF, Xiang X, Liu Y, Kang X, Song Y, Guo X, Liu H, Ding N, Zhang T, Duan P, Lin Y, Zheng W, Wang X, Lin N, Tu M, Xie Y, Zhang C, Liu W, Deng L, Gao S, Ping L, Wang X, Zhou N, Zhang J, Wang Y, Lin S, Mamuti M, Yu X, Fang L, Wang S, Song H, Wang G, Jones L, Zhu J, Chen SY. A safe and potent anti-CD19 CAR T cell therapy. Nat Med. 2019 Jun;25(6):947-953. doi: 10.1038/s41591-019-0421-7. Epub 2019 Apr 22. PMID 31011207